CLINICAL TRIAL: NCT04398914
Title: A Randomised, Multicenter, Open-label, Phase II Study Evaluating Pyrotinib Plus Trastuzumab, Pertuzumab and Nab-paclitaxel as Neoadjuvant Therapy in Early Stage or Locally Advanced Human Epidermal Growth Factor Receptor (HER) 2 - Positive Breast Cancer
Brief Title: Pyrotinib, Trastuzumab, Pertuzumab and Nab-paclitaxel as Neoadjuvant Therapy in HER2-positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJBC2001
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer Invasive
Keywords: HER2-positive; Stage II-III
MeSH Terms: interventions — pyrotinib; Trastuzumab; pertuzumab; 130-nm albumin-bound paclitaxel; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyrotinib, trastuzumab, pertuzmab and paclitaxel (Experimental): Prior to surgery: pyrotinib, trastuzumab, pertuzumab and nab-paclitaxel for 4 cycles (1 cycle = 21 days).
  After surgery：
  * if non-tpCR：chemotherapy with epirubicin and cyclophosphamide (EC), followed with pertuzumab and trastuzumab up to 1 year total; or T-DM1 for 14 cycles.
  * if tpCR: chemotherapy 0-4 cycles according to physician's choice, followed with pertuzumab and trastuzumab up to 1 year total.
  Interventions: Drug: Pyrotinib; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Nab-paclitaxel; Drug: EC chemotherapy; Drug: Physician's choice; Drug: T-DM1; Procedure: Surgery
- Trastuzumab, pertuzmab and paclitaxel (Active Comparator): Prior to surgery: trastuzumab, pertuzumab and nab-paclitaxel for 4 cycles (1 cycle = 21 days).
  After surgery：
  * if non-tpCR：chemotherapy with epirubicin and cyclophosphamide (EC), followed with pertuzumab and trastuzumab up to 1 year total; or T-DM1 for 14 cycles.
  * if tpCR: chemotherapy 0-4 cycles according to physician's choice; followed with pertuzumab and trastuzumab up to 1 year total.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Nab-paclitaxel; Drug: EC chemotherapy; Drug: Physician's choice; Drug: T-DM1; Procedure: Surgery

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib 400 mg taken orally everyday, every 3 weeks, for 4 cycles.
  Arms: Pyrotinib, trastuzumab, pertuzmab and paclitaxel
Drug: Trastuzumab — Trastuzumab IV infusion in 3-week cycles.
  Neoadjuvant treatment: 8 milligrams per kilogram (mg/kg) loading dose for Cycle 1, followed by 6 mg/kg for Cycles 2-4.
  Adjuvant treatment: 8 mg/kg loading dose, followed by 6 mg/kg for remaining cycles till completion of 1 year trastuzumab
Drug: Pertuzumab — Pertuzumab IV infusion in 3-week cycles.
  Neoadjuvant treatment: 840 milligrams (mg) loading dose for Cycle 1, followed by 420 mg for Cycles 2-4.
  Adjuvant treatment: 840 mg loading dose, followed by 420mg for remaining cycles till completion of 1 year pertuzumab
Drug: Nab-paclitaxel — Nab-paclitaxel 100mg/m2 by intravenous (IV) infusion on day1, day8 and day15, every 3 weeks, for 4 cycles.
Drug: EC chemotherapy — Epirubicin 90 mg/m2, and cyclophosphamide 600 mg/m2 by intravenous (IV) infusion every 3 weeks for 4 cycles (Cycles 5-8)
Drug: Physician's choice — Physician decided chemotherapy for 0-4 cycles.
Drug: T-DM1 — T-DM1 IV infusion in 3-week cycles. 3.6 mg/kg by intravenous (IV) infusion every 3 weeks for 14 cycles
Procedure: Surgery — All participants who are eligible for surgery will undergo surgery and have their pathologic response evaluated.

SUMMARY:
This study aims to evaluate the efficacy and safety of pyrotinib in combination with trastuzumab, pertuzumab and nab-paclitaxel as neoadjuvant therapy in early stage or locally advanced HER2-positive breast cancer.

DETAILED DESCRIPTION:
The study evaluate the pathological complete response rate, event-free survival, disease-free survival, overall survival and safety of pyrotinib in combination with trastuzumab, pertuzumab and nab-paclitaxel as neoadjuvant therapy in early stage or locally advanced HER2-positive breast cancer. Patients will receive 4 cycles of pyrotinib in combination with trastuzumab, pertuzumab and nab-paclitaxel or 4 cycles of trastuzumab, pertuzumab and nab-paclitaxel as neoadjuvant therapy, then undergo surgery, then receive adjuvant chemotherapy and targeted therapy according to pathologic response and physician's choice.

ELIGIBILITY:
Inclusion Criteria:

* With signed consent
* Histologically confirmed invasive breast carcinoma with a primary tumor size of no less than (≥) 2 centimeters (cm) by standard local assessment technique
* Breast cancer stage at presentation: stage II-III
* HER2-positive breast cancer defined as 3+ score by immunohistochemistry in > 10 percent (%) of immunoreactive cells or HER2 gene amplification by in situ hybridization
* Known hormone receptor status (estrogen receptor and/or progesterone receptor)
* Eastern Cooperative Oncology Group Performance Status equal to or less than (<=) 1
* Baseline left ventricular ejection fracture >= 50% measured by echocardiography
* Willing to use highly effective form of nonhormonal contraception while on study and for 7 months after end of study treatment for female with fertility or male
* Willing to obey the study protocol

Exclusion Criteria:

* Stage IV disease
* Previous anti-cancer therapy or radiotherapy for any malignancy
* History of other malignancy within 5 years prior to screening, except for appropriately-treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, ,Stage I uterine cancer or thyroid papillary microcarcinoma
* Concurrent anti-cancer treatment in another investigational trial, including hormone therapy, bisphosphonate therapy, or immunotherapy
* Major surgical procedure unrelated to breast cancer within 4 weeks prior to randomization or from which the participant has not fully recovered
* Serious cardiac illness or medical condition
* Other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness
* Any abnormalities in liver, kidney or hematologic function laboratory tests immediately prior to randomization
* Sensitivity to any of the study medications, any of the ingredients or excipients of these medications, or benzyl alcohol
* Not able to swallow the drug
* Pregnant or lactating
* Positive serum or urine pregnancy test or above mentioned tests cannot be achieved for women with fertility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Total Pathologic Complete Response (tpCR) | After completion of 4 cycles of neoadjuvant therapy. The duration of one treatment cycle is 21 days
  tpCR is defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes after completion of neoadjuvant therapy and surgery (that is, ypT0/is, ypN0, in accordance with the current American Joint Committee on Cancer [AJCC] staging system).The duration of one treatment cycle is 21 days.

SECONDARY OUTCOMES:
Percentage of Participants With Breast Pathologic Complete Response (bpCR) | After completion of 4 cycles of neoadjuvant therapy The duration of one treatment cycle is 21 days. at the time of surgery
  bpCR is defined as the absence of any residual invasive cancer on the hematoxylin and eosin evaluation of the resected breast specimen after completion of neoadjuvant therapy and surgery (that is, ypT0/is, in accordance with current AJCC staging system).The duration of one treatment cycle is 21 days.
Clinical response | Cycle 1-4. The duration of one treatment cycle is 21 days.
  Percentage of Participants With Complete Response, Partial Response, Stable Disease, or Progressive Disease During Cycles 1-4, According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. The duration of one treatment cycle is 21 days.
Event-free survival (EFS) | From Baseline to EFS event or date last known to be alive and event-free (up to 5 years)
  EFS is defined as the time from randomization to the first documentation of one of the following events: Disease progression (before surgery) as determined by the investigator with use of RECIST v1.1 Any evidence of contralateral disease in situ was not identified as progressive disease; Disease recurrence (local, regional, distant, or contralateral) after surgery; Death from any cause.
Disease-free survival (DFS) | From surgery to DFS event or date last known to be alive and event-free (up to 5 years)
  DFS was defined as the time from first date of no disease (i.e., date of surgery) to first documentation of one of the following events: Disease recurrence (local, regional, distant, or contralateral) after surgery. Any evidence of contralateral disease in situ was not identified as disease recurrence; Death from any cause.
Overall survival (OS) | From Baseline to OS event or date last known to be alive (up to 5 years)
  OS was defined as the time from randomization to death from any cause.

OTHER OUTCOMES:
Percentage of Participants With At Least One Adverse Event During Treatment Period | From randomization to 30 days after completion of study treatment
  The percentage of participants who experienced at least one adverse event during the neoadjuvant period, surgery, adjuvant treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Kunwei Shen, MD,PhD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No